CLINICAL TRIAL: NCT02744001
Title: Diet Study: The Reinforcing Value of Added Sugars
Brief Title: The Reinforcing Value of Added Sugars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GFHNRC148
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Added Sugar Diet (Experimental): Menu containing <10% of total daily energy intake from added sugars.
  Interventions: Other: Low Added Sugar Diet

INTERVENTIONS:
Other: Low Added Sugar Diet — 1-week intake of Low Added Sugar Diet 3 day rotating menu

SUMMARY:
The purpose of this study is to determine how daily diet relates to eating choices.

DETAILED DESCRIPTION:
Despite the long-term emphasis on reducing intake of and added sugar, this behavioral change has been hard to instill amongst most of the population. Foods with added sugars are highly reinforcing and, as such, reducing their consumption in order to adhere to the dietary guidelines (DGA) may be difficult to maintain. Sugar produces effects similar to some drugs of abuse such as increased extracellular dopamine release in the nucleus accumbens shell resulting in a reinforcing effect. Reducing any reinforcing behavior can be challenging, but in terms of food, it is not known whether the reinforcing value of foods high in added sugar increases when access to these foods is reduced. If so, this would present a mechanistic barrier to meeting the DGA and making dietary changes in general. That the reinforcing value of a behavior (e.g., eating sugar) will be increased when the rate of that behavior is decreased has strong theoretical underpinnings in the "Disequilibrium Approach". This theory predicts that the circumstances of reinforcement are created or limited by changing baseline access. According to the Disequilibrium Approach, a response deficit will result in an increase in reinforcement. Applied to the proposed study, the Disequilibrium Approach would predict that lowering the consumption of dietary added sugar would increase the reinforcing value of foods high in added sugar. The Disequilibrium Approach has accurately predicted an increase in the relative reinforcing value (RRV) of snack foods among children. However, dietary changes would need to occur at the whole diet level for adults and children to meet the DGA for reducing added sugar intake. It is important to know if reducing added sugars at the whole-diet level results in increases in the reinforcing value of foods high in added sugars.

ELIGIBILITY:
Inclusion Criteria:

* BMI within 18.5-24.9 kg/m2 or BMI within 30.0-50.0 kg/m2
* Willing to consent to study conditions
* Habitually consume at least 10% of daily energy intake from added sugars

Exclusion Criteria:

* BMI 25.0-29.9 kg/m2
* Currently taking drugs that change hunger
* Have an eating disorder
* Current tobacco user
* Have diabetes or heart disease
* Pregnant, lactating or planning pregnancy
* Low liking of all available study test foods
* Allergy/aversion to any of the foods provided during the diet intervention

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Change in relative reinforcing value (RRV) of snacks as assessed by indicator | Baseline and 1 week
  RRV of snacks will be assessed by evaluating the number of responses (mouse button presses) a subject is willing to complete to gain access to a high added sugar snack or low added sugar alternative.

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flack KD, Ufholz K, Casperson S, Jahns L, Johnson L, Roemmich JN. Decreasing the Consumption of Foods with Sugar Increases Their Reinforcing Value: A Potential Barrier for Dietary Behavior Change. J Acad Nutr Diet. 2019 Jul;119(7):1099-1108. doi: 10.1016/j.jand.2018.12.016. Epub 2019 Apr 6. PMID 30962120